CLINICAL TRIAL: NCT06245915
Title: An Open-label, Multicenter Phase 1/2 Study to Evaluate the Safety and Efficacy of AB-2100 in Patients With Recurrent Advanced or Metastatic Clear-cell Renal Cell Carcinoma (ccRCC)
Brief Title: AB-2100, an Integrated Circuit T Cell Therapy in Patients With Recurrent Clear-cell Renal Cell Carcinoma (ccRCC)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arsenal Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AB-2100-201
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Advanced/Metastatic Clear Cell Renal Cell Carcinoma; Recurrence
Keywords: kidney cancer; CAR T; Cell Therapy; Autologous; Autologous Cell Therapy; ccRCC; Clear Cell Renal Cell Carcinoma; AB-2100; Integrated Circuit T Cell
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma; Recurrence; Kidney Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AB-2100 (Experimental): Patients receive a single dose of AB-2100 intravenously on day 0. Patients may be assigned to receive conditioning chemotherapy prior to the infusion.
  Interventions: Biological: AB-2100

INTERVENTIONS:
Biological: AB-2100 — autologous T cell therapy
  Other Names: Integrated Circuit T cells

SUMMARY:
This is a multi-center, open-label phase 1/2 trial evaluating the safety and efficacy of AB-2100 cell product. The study may enroll approximately 60 patients in phase 1 and approximately 70 patients in phase 2.

DETAILED DESCRIPTION:
This study is intended for the patients who have been diagnosed with clear-cell renal cell carcinoma that either came back or did not improve after treatment with a checkpoint inhibitor and a VEGF inhibitor. The purpose of this study is to test the safety and efficacy of AB-2100 cells in patients with renal cell carcinoma. This treatment has not been approved by the Food and Drug Administration.

The goal of this study is to determine the maximum tolerated dose of the AB-2100 cells. T cells are part of the immune system that protect the body from infection and may help fight cancer. The T cells given in this study will come from the patient and will have a genetic circuit/logic gate put in them that makes them able to recognize prostate-specific membrane antigen (PSMA) and carbonic anhydrase 9 (CA9), 2 proteins found on tumor cells. These logic-gated T cells may help the body's immune system identify and kill cancer cells while sparing normal healthy tissues from toxicity.

The AB-2100 cells are given as a single intravenous infusion. Patients may be assigned to receive conditioning chemotherapy prior to the infusion

After completion of study treatment, patients are followed with serial measurements of safety, tolerability and response.

This is a research study to obtain new information that may help people in the future.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or metastatic clear-cell renal cell carcinoma
* Must have received an immune checkpoint inhibitor and a VEGF-targeted therapy in the advanced or metastatic setting. Must have evidence of progression on or after the last treatment regimen or discontinued treatment for unacceptable toxicity.
* Adequate organ function as per protocol definitions.
* Eastern Cooperative Oncology Group (ECOG) performance status score 0 or 1.
* Measurable disease at time of enrollment as per protocol definitions.
* Female subjects of childbearing potential and male subjects must agree to use acceptable method(s) of contraception from enrollment through at least 12 months after AB-2100 infusion.

Exclusion Criteria:

* Any prior systemic RCC therapy within 14 days of time of cell collection (interval of 28 days will be required if the last immediate treatment contained an antibody-based agent).
* Systemic anti-cancer therapy within 14 days of starting of conditioning chemotherapy (interval of 28 days will be required if the last immediate treatment contained an antibody-based agent)
* Investigational cellular therapies within 8 weeks prior to start of conditioning chemotherapy
* Prior treatment with anti-CA9 therapies
* Myocardial infarction or unstable angina within 6 months prior to screening
* Pleural effusion that requires drainage for symptom management within 28 days of screening.
* Active autoimmune disease requiring immunosuppressive therapy or uncontrolled with treatment.
* Untreated brain metastasis.
* Subjects unwilling to participate in an extended safety monitoring period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1 (Dose escalation): incidence of adverse events | From AB-2100 infusion up to 21 days post infusion
  Defined as dose-limiting toxicities based on a 3+3 dose escalation study design
Phase 2 (Cohort expansion): Objective response rate (ORR) | From AB-2100 infusion up to 24 months post-infusion
  ORR based on Independent Review Committee (IRC) assessment, defined as the proportion of subjects who have achieved a best overall response of CR or PR according to RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Arsenal Biosciences, Study Director — Arsenal Biosciences
Locations (9):
- United States (9):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - City of Hope, Duarte, California
  - Moffitt Cancer Center, Tampa, Florida
  - University of Iowa and Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Dana Farber Cancer Institue, Boston, Massachusetts
  - Perlmutter Cancer Center - NYU Langone Health, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute - Univ of Utah Health, Salt Lake City, Utah